CLINICAL TRIAL: NCT06872931
Title: Investigation of the Effects of C-Mill (Hocoma AG, Switzerland) Treadmill Training on Trunk Balance in Patients with Spinal Cord Injury
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Sinem Yıldırım, MSc Physiotherapist, Ankara City Hospital Bilkent
Other Study IDs: TABED 1-24-346
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Postural balance
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- conventional balance exercises: In addition to conventional therapy, conventional balance exercises group will undergo conventional balance exercises and gait training, either within or outside the parallel bars, for a minimum of two days per week in 30-minute sessions. Over four weeks, they will complete a total of 10 sessions of gait and balance training.
- Treadmill training group: In addition to conventional therapy, the Treadmill training group will undergo static and dynamic balance exercises and gait training on the C-Mill platform for a minimum of two days per week, with sessions lasting 30 minutes each. Over four weeks, they will complete a total of 10 sessions of gait and balance training on the C-Mill platform.

SUMMARY:
This study examines how C-Mill treadmill training affects balance and stability in people with spinal cord injury (SCI). Many individuals with SCI experience difficulty with sitting and walking balance, which affects their daily activities and independence. This research aims to explore whether C-Mill, a treadmill that combines virtual reality and sensor-based walking support, can improve trunk stability and mobility.

Who Can Join the Study?

People who:

Are between 18-65 years old Have a spinal cord injury at T4 or lower Are classified as ASIA C or D (moderate to mild impairment) Have stable spinal alignment and can safely participate in walking exercises People who have osteoporosis, heart or lung conditions, additional neurological diseases, or severe joint problems cannot participate.

Our study is a prospective observational study. Regardless of whether exercises are performed conventionally or on an alternative gait platform such as the C-Mill, all interventions are part of routine clinical practice. Patients whose treatment programs already align with the aforementioned procedures will be included. In robotic rehabilitation and assisted gait device laboratories equipped with the C-Mill platform, spinal cord injury patients follow a standardized rehabilitation protocol. These laboratories operate on an appointment-based system. After random group allocation, patients in the study group will undergo assessments at the beginning and end of C-Mill therapy, while control group patients will be enrolled before initiating C-Mill treatment. Following data collection for the control group, these patients will also receive C-Mill therapy.

What Will Happen in the Study?

Participants will be randomly assigned to one of two groups:

C-Mill Group: Receives standard rehabilitation plus C-Mill treadmill training for balance and walking exercises (10 sessions over 4 weeks).

Conventional Therapy Group: Receives standard rehabilitation plus traditional balance and walking exercises (10 sessions over 4 weeks).

How Will the Results Be Measured?

Researchers will assess:

Balance and Stability using functional reach and trunk control tests Independence in Daily Life using a spinal cord-specific scale (SCIM-III) Quality of Life using a health questionnaire (SF-36) Fear of Falling using a visual scale Why Is This Study Important? The study aims to determine if C-Mill training is more effective than traditional rehabilitation in improving balance, stability, and confidence in movement for people with SCI.

DETAILED DESCRIPTION:
Enhancing trunk balance and stability is a key objective in SCI rehabilitation. Various exercise modalities, including proprioceptive training, core strengthening, yoga, and Pilates, are employed to improve motor skills, coordination, and quality of life. Recently, virtual reality (VR)-based approaches, such as the C-Mill treadmill (Hocoma AG, Switzerland), have gained prominence. The C-Mill integrates visual and motor training through a suspension-supported system that ensures safe ambulation while adapting to the patient's pace. Unlike conventional treadmills and robotic-assisted devices, it uniquely incorporates VR to simulate real-world gait challenges, bridging the gap between traditional therapies and independent walking.

This study aims to investigate the effects of gait exercises performed with the C-Mill treadmill on trunk balance and stability by leveraging its advantages, such as gradual weight-bearing, improved gait stability, and reduced fatigue.

Our study is a prospective observational study. Regardless of whether exercises are performed conventionally or on an alternative gait platform such as the C-Mill, all interventions are part of routine clinical practice. Patients whose treatment programs already align with the aforementioned procedures will be included. In robotic rehabilitation and assisted gait device laboratories equipped with the C-Mill platform, spinal cord injury patients follow a standardized rehabilitation protocol. These laboratories operate on an appointment-based system. After random group allocation, patients in the study group will undergo assessments at the beginning and end of C-Mill therapy, while control group patients will be enrolled before initiating C-Mill treatment. Following data collection for the control group, these patients will also receive C-Mill therapy. The study aims to identify differences in outcomes between the applied interventions.

Data Quality and Management Procedures Patients admitted for inpatient treatment at the Spinal Cord Injury Rehabilitation Clinic of Ankara Bilkent City Hospital, who meet the inclusion criteria and voluntarily agree to participate in the study by reading and signing the informed consent form, will be included in the study. The medical status of all participants will be evaluated and recorded by the clinical research responsible physician.

A predefined data management plan will be implemented for missing, inconsistent, or erroneous data. Missing data will be identified and analyzed using statistical methods such as multiple imputation when necessary.

To ensure the integrity of data entry, regular audits and consistency checks will be performed by a physiotherapist involved in the study. To increase the reliability of the data, patient records and assessment reports will be cross-checked with the collected data. This will include comparisons made with electronic health records, paper-based case reports, and direct observation notes. All study procedures, including patient recruitment, data collection, data entry, data analysis, and reporting of adverse events, will be carried out according to predefined criteria.

Any adverse events or unexpected complications occurring during the study will be systematically documented and reported.

The determination of the appropriate sample size was based on the study by Khurana et al. A priori power analysis was conducted using the G* Power software (version 3.0.10, Universität Düsseldorf, Düsseldorf, Germany). The sample size for our study was calculated to include a minimum of 11 patients per group, ensuring 80% power with an alpha error rate of 0.05.

For statistical analysis, descriptive statistics will be presented as the mean and standard deviation for numerical variables if the parametric assumptions are met, and as the median and minimum-maximum values if the parametric assumptions are not met. For categorical variables, frequency and percentage values will be reported. The statistical significance of differences between groups will be examined using the Independent Samples T-Test if parametric assumptions are met, and the Mann-Whitney U Test if parametric assumptions are not met. Analyses will be conducted with a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* SCI at T4 or below
* ASIA classification C or D
* Spinal stabilization achieved
* Willingness to participate voluntarily

Exclusion Criteria:

* Osteoporosis
* Cardiopulmonary disease
* Neurological conditions other than SCI
* Joint or musculoskeletal disorders
* Presence of orthostatic hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be treated at Ankara City Hospital, Department of Physical Medicine and Rehabilitation, within the Neurophysiological Exercise and Robotic Rehabilitation Laboratories.
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
Functional Reach Test | Four weeks
  The patient is instructed to stand next to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist.
  The assessor records the starting position at the 3rd metacarpal head on the yardstick.
  Patient is instructed to reach as farther as possible without moving from the ground The location of the 3rd metacarpal is recorded again. Scores are determined by assessing the difference between the start and end position is the reach distance, usually measured in inches.
  Three trials are done and the average of the last two is noted

SECONDARY OUTCOMES:
Berg Balance Scale | Four weeks
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
36-Item Short Form Survey (SF-36) | Four weeks
  SF-36 Short Form will be used to assess quality of life. This questionnaire consists of 36 questions and 8 sub-parameters in total. Sub-parameters are determined as physical function, physical role difficulty, pain, general health, vitality, social function, emotional role function and mental health. It is in the form of a scale with points from zero (worst health) to 100 (best health status).
Spinal Cord Independence Measure (SCIM) | Four weeks
  The SCIM has been developed to address three specific areas of function in patients with spinal cord injuries (SCI). It looks at self-care (feeding, grooming, bathing, and dressing), respiration and sphincter management, and a patient's mobility abilities (bed and transfers and indoors/outdoors). A clinician or member of the clinical staff scores the patient on the items that this outcome measure addresses. Its scoring system is self-explanatory; therefore there isn't a manual to instruct the clinician in the scoring process. Scores range from 0-100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence. Each subscale score is evaluated within the 100-point scale (self-care: 0-20; respiration and sphincter management: 0-40; mobility: 0-40).
Trunk Stability Measurement | Four weeks
  Trunk Stability assessment will be performed using the HUR Smart Balance® (HUR International, FINLAND) device. The HUR Smart Balance System® consists of a BTG4-FE platform, All-in-One Computer, Balance Support Station and HUR Smart Balance Software. The platform will be checked before each test. The analysis will be performed with the patient standing on the platform, barefoot, 2 cm between heels, arms on both sides of the body. At least 5 seconds (preliminary phase) will be immobile before starting the assessment. After the preliminary phase, patients will stand in an upright position with their arms at their sides. The analysis duration will be 60 seconds. Postural sway and balance parameters will be measured in the static balance test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No